CLINICAL TRIAL: NCT07005622
Title: Inspiratory Muscle Training Using the O2 Trainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sam Houston State University (Other)
Responsible Party: Principal Investigator, Patrick Davis, Director of Research, Sam Houston State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2024-116
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Inspiratory Muscle Training; Blood Pressure
Keywords: Maximal Respiratory Pressures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will practice deep breathing exercise 5 times per week
  Interventions: Other: Deep breathing
- Experimental Group (Experimental): The experimental group will participate in inspiratory muscle training 5 times per week
  Interventions: Other: O2 Trainer

INTERVENTIONS:
Other: O2 Trainer — The O2 Trainer uses varying caps to limit airflow during inspiration.
  Arms: Experimental Group
Other: Deep breathing — Comparator/placebo for the control group
  Arms: Control Group

SUMMARY:
This study aims to investigate the effects of resistive inspiratory training using the O2 Trainer on cardiopulmonary outcomes in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Able to participate in training 5 days per week

Exclusion Criteria:

* Previous ventilation
* Diagnosed chronic obstructive pulmonary disease (COPD)
* Uncontrolled asthma
* Previous ear drum rupture
* Previous abdominal hernia
* Acute respiratory infection
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Force | Change following 5-6 weeks of training
  Inspiratory force (mmHg) will be measured using a digital pressure gauge connected to a mouthpiece.

SECONDARY OUTCOMES:
Blood Pressure | Change following 5-6 weeks of training
  mmHG measured by FDA approved automated blood pressure cuff.
Resting Heart Rate | Change following 5-6 weeks of training
  Beats per minute, measured using a chest worn heart rate monitor.
Heart Rate Variability | Change following 5-6 weeks of training
  Measured using a chest worn heart rate monitor.
Diaphragm Thickness | Change following 5-6 weeks of training
  Measured by ultrasound

OTHER OUTCOMES:
Handgrip strength via handgrip dynamometer | Change following 5-6 weeks of training
  Strength of handgrip will be recorded as kg of force using a handgrip dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sam Houston State University College of Osteopathic Medicine, Conroe, Texas, United States

IPD SHARING:
Plan to Share IPD: No